CLINICAL TRIAL: NCT01850121
Title: Remicade in the Treatment of Patients With Active Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Helena Forsblad d'Elia, MD, PhD, Göteborg University
Other Study IDs: 2002-11-04 amended 2002-01-08
Record Dates: First submitted 2013-05-06; First posted 2013-05-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; infiximab; single armed trial
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab: Patients with active AS defined as BASDAI score above 4 and no exclusion criteria were consecutively included in this single-armed unblinded trial.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — 5 mg/kg every 6 weeks during the first year and 3 mg/kg every 8 weeks during the second year. Concomitant treatment with methotrexate 7.5 mg/week.
  Other Names: Remicade

SUMMARY:
The aim of the study was to evaluate the efficacy of infliximab (IFX) treatment, 5 mg/kg every 6 weeks, in patients with active ankylosing spondylitis (AS) and to determine whether IFX dose reduction and interval extension, 3 mg/kg every 8 weeks during the second year sustained the treatment effect. The study was started in 2003 an finished in 2008.

ELIGIBILITY:
Inclusion Criteria:

The patients had to fulfill the following four inclusion criteria:

(I) Age between 18 and 60 years, (II) proven diagnosis according to the modified New York criteria 12 for definitive AS, (III) active disease with Bath AS Disease Activity Index (BASDAI) score above 4 and (IV) current or previous treatment with conventional non-steroidal anti-inflammatory drugs (NSAID) in adequate doses without sufficient effect.

Exclusion Criteria:

* current signs or symptoms of severe, progressive or uncontrolled hepatic, hematological, pulmonary, cardiac, neurological or cerebral disease;
* ongoing or past serious infection (including HIV and past or current tuberculosis);
* pregnancy or breast feeding;
* current malignancy or history of malignancy within the past five years;
* congestive heart failure and any contraindication to MRI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with active ankylosing spondylitis with BASDAI>4
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2003-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Bath AS disease activity score (BASDAI) | 16 weeks
  The proportion of responders at week 16 defined as a reduction of 50% and/or 2 units improvement from baseline of Bath AS disease activity score (BASDAI)

CONTACTS AND LOCATIONS:
Overall Officials: Boel Morck, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Morck B, Pullerits R, Geijer M, Bremell T, Forsblad-d'Elia H. Infliximab dose reduction sustains the clinical treatment effect in active HLAB27 positive ankylosing spondylitis: a two-year pilot study. Mediators Inflamm. 2013;2013:289845. doi: 10.1155/2013/289845. Epub 2013 Sep 5. PMID 24089587